CLINICAL TRIAL: NCT06520020
Title: Evaluating Safety and Feasibility of Transcutaneous Spinal Cord Stimulation Following Traumatic and Non-Traumatic Spinal Cord Injury: A Pilot Study
Acronym: STIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Francis Farhadi (Other)
Responsible Party: Sponsor-Investigator, Francis Farhadi, Associate Professor, Neurosurgery, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 96620
Record Dates: First submitted 2024-07-11; First posted 2024-07-25 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Spinal Cord Stimulation; Electric Stimulation Therapy; Traumatic Spinal Cord Injury; Cervical Myelopathy
Keywords: Stimulation; Transcutaneous; MagStim; Transcranial; Magnetic
MeSH Terms: interventions — Electric Stimulation

STUDY DESIGN:
Intervention Model Description: The study will be a non-randomized, non-blinded pilot study to analyze the safety and feasibility of a non-significant risk device, using transcutaneous spinal cord stimulation.
  We aim to include 30 total patients, 10 patients in each of 3 groups:
  1. Non-traumatic spinal cord injury (ntSCI) with diagnosis of degenerative cervical myelopathy and offered surgical intervention.
  2. Early tSCI screened during the hospital admission when cervical/thoracic spinal injury was diagnosed.
  3. Delayed tSCI (control) screened 6-24 months after acute cervical/thoracic spinal injury.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Non-Traumatic Spinal Cord Injury (ntSCI,) DCM - Progressive (Experimental): Non-traumatic spinal cord injury (ntSCI) with diagnosis of degenerative cervical myelopathy (DCM) and offered surgical intervention. Prospective.
  Interventions: Device: Transcutaneous Spinal Cord Stimulation (Tc-SCS)
- Traumatic Spinal Cord Injury (tSCI) - Early/Acute (Experimental): Traumatic spinal cord injury (tSCI) screened during the hospital admission when cervical/thoracic spinal injury was diagnosed. 2-6 weeks after injury.
  Interventions: Device: Transcutaneous Spinal Cord Stimulation (Tc-SCS)
- Traumatic Spinal Cord Injury (tSCI) - Chronic (Active Comparator): Delayed traumatic spinal cord injury (tSCI) screened 6-24 months after acute cervical/thoracic spinal injury. The use of transcutaneous spinal cord stimulation (Tc-SCS) in chronic SCI delivered in the delayed timeframe is relatively well studied, and therefore will serve as the control arm.
  Interventions: Device: Transcutaneous Spinal Cord Stimulation (Tc-SCS)

INTERVENTIONS:
Device: Transcutaneous Spinal Cord Stimulation (Tc-SCS) — This study will employ a DS8R Biphasic Constant Current Stimulator (Digitimer, Hertfordshire, United Kingdom) to administer transcutaneous (Tc) SCS through bursts of biphasic rectangular pulses, each lasting 400 μs to 1 ms, at 30 Hz frequency on a carrier frequency is 10 kHz. The intensity of stimulation will be 120% the threshold intensity that elicits visible twitch or motor evoked potential (MEP) triggered in the biceps brachii (BB) or abductor pollicis brevis (APB) muscle for upper extremity, and quadriceps femoris (QF) or tibialis anterior (TA) in the lower extremity.
  Other Names: Electrical Stimulation

SUMMARY:
The study will be a non-randomized, non-blinded pilot study to analyze the safety and feasibility of a non-significant risk device, transcutaneous spinal cord stimulation. The aim is to include 30 total patients, 10 patients in each of 3 groups:

1. Non-traumatic spinal cord injury (ntSCI) with diagnosis of degenerative cervical myelopathy and offered surgical intervention.
2. Early tSCI screened during the hospital admission when cervical/thoracic spinal injury was diagnosed.
3. Delayed tSCI (control) screened 6-24 months after acute cervical/thoracic spinal injury.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) can result from primary physical insults such as acute trauma, or secondary insults that result from chronic compression and ischemia. The resultant neurological impairment leads to high personal and societal burden. There are few effective therapies to improve function for those living with SCI. Spinal cord stimulation (SCS) represents a safe and potentially effective treatment for persons with SCI-related pain and paralysis. The aim of this study is to investigate the potential clinical utility of SCS delivered transcutaneously in patients at various stages of SCI, resulting from traumatic and non-traumatic mechanisms. This study will evaluate the ability to safely stimulate the injured spinal cord at defined intervals and record autonomic and sensorimotor function of participants across their admission, rehabilitation, and clinical follow-up.

Various upper and lower extremity-related functional measures will be assessed at baseline and at established follow-up timepoints across a 12-month period. The safety of this intervention, and the utility of each outcome measure will be the primary outcome of the study. To our knowledge, there are no reported clinical trials that have evaluated multi-modal outcomes of SCS. Furthermore, there are no proposed trials of SCS for these SCI subtypes across the post-injury spectrum posted to the platform clinicaltrials.gov. Data obtained from this pilot evaluation will be used to inform an early phase Ib/II trial of efficacy for improvement of paralysis, autonomic dysfunction, and pain following SCI.

Over 2.5 million Americans are living with various forms of SCI, equating to substantial individual and societal burden (1). Acute traumatic SCI average costs alone range from $380K to $1.4M. This high socioeconomic impact has undergone significant inflation with estimated annual costs of $4 billion in 1990, recently increasing to $23 billion. Approximately 13,000 new traumatic SCI events are noted yearly in North America. Degenerative cervical myelopathy (DCM) represents the most prevalent etiology of nontraumatic spinal cord (ntSCI) and dysfunction in adults. The prevalence of ntSCI is order(s) of magnitude higher than that of tSCI.

Together, these conditions significantly impact millions of North Americans often with greater personal impact that chronic conditions such as diabetes or cardiac disease. The considerable societal concern due to this individual disability is compounded by the lack of viable treatment options.

DCM arises from age-related degenerative processes, leading to osteophyte development, facet joint enlargement, ossification of spinal ligaments, and disk protrusion. These arthritic changes collectively compress the spinal cord causing injury with associated ischemia and inflammation. In turn, a similar constellation of symptoms develop including extremity pain, reduced motor function, numbness, hemodynamic lability, urinary incontinence, bowel dysfunction, and walking instability contributing towards higher years lived with disability (DALYs) as well as overall economic burden.

Currently, effective evidence-proven treatments are restricted to surgical decompression and rehabilitation. Narrative studies have shown that patients living with paralysis want options for neural modulation therapies, as they perceive the risk-to-benefit ratio of implanted devices more favorably than healthcare professionals. Given overall suboptimal outcomes in patients with SCI, it is critical to further enhance both the recovery rates and the extent of recovery beyond what is achievable through surgical decompression.

Spinal cord stimulation has been shown to mediate functional improvement following acute traumatic SCI in terms of limb function, ambulation, hand strength, autonomic dysfunction, intractable pain, and bladder control. The majority of published studies have applied stimulation during the chronic phase of recovery, and largely in a single or small group of participants.

Variable applications of SCS for SCI have yet to be demonstrated using multi-modality stimulation, such as spinal transcutaneous, spinal epidural, and transcranial magnetic stimulation of the motor cortex. Harkema and colleagues demonstrated that epidural SCS can return volitional motor control in participants who had none following chronic thoracic injury. Their work at the University of Louisville also has shown that multilevel transcutaneous spinal cord stimulation can be applied to several cervicothoracic regions spanning across the entire limb enlargement, and provide sensorimotor functional improvements during neurorehabilitation. These approaches have subsequently been applied at other centers with success for sensorimotor recovery.

The utilization of SCS in managing Failed Back Surgery Syndrome (FBSS), Complex Regional Pain Syndrome (CRPS), and chronic leg ischemia has been well documented. However, there is limited evidence indicating the use of SCS in patients with tSCI or ntSCI with regards to improving motor functions. This application of SCS could identify important differentiators in neural modulation that will correspond to improved functional outcomes, patient reported outcome measures (PROM), and quality of life (QoL). Should differentiators be observed, these conclusions will inform phase Ib/II study of SCS-based neuromodulation vs standard-of-care rehabilitation. This is directly in line with the best-of-practice and goals promoted by the leaders in SCI clinical research and patient-driven goals.

To date, there are no reported clinical trials involving participants in the subacute phase of tSCI, despite the widely-held belief that this phase offers the greatest potential for therapeutic intervention to reduce secondary injury and preserve functional networks.

Likewise, there are no clinical trials examining the role of perioperative SCS in patients diagnosed with any form of ntSCI (including patients with DCM who undergo surgical decompression).

The proposed study will directly address whether neuromodulation has a specific therapeutic potential for persons having sustained acute traumatic and non-traumatic spinal injuries. This study will specifically address whether this can be achieved with a non-significant risk device such as transcutaneous spinal cord stimulation. Lastly, this study will comparatively assess the modalities that can be used to reliably stimulate and measure the physiologic effects of neuromodulation of the injured spinal cord.

Additionally, this study aims to test the hypothesis that transcutaneous electrical spinal cord stimulation has equivalent modulatory effect on sensorimotor pathways and spinal cord function. This study will prospectively record neurologic outcomes to fully leverage the technologies at our disposal and maximize the potential benefit for each participant. The subsequent results will further help determine whether spinal cord neuromodulation can be directly correlated to either patient reported outcome or functional performance measures. Moreover, to determine feasibility of transcutaneous SCS at various timepoints after presentation, this study will measure spinal signal outputs before and after standard-of-care treatments including surgery and intensive neural rehabilitation.

The preliminary data in support of SCS for individuals with tSCI applied at chronic recovery phases has demonstrated promising outcomes, potentially ameliorating this severe condition. The investigation into utilizing SCS as a management approach for acute tSCI and ntSCI (ie. DCM), in conjunction with surgical interventions and rehabilitation, represents a promising prospect for enhancing the quality of life of those afflicted with this debilitating neurological disorder.

ELIGIBILITY:
Inclusion Criteria:

* Age: = 18 years and = 80 years.
* Written informed consent by patient and/or legal authorized representative (LAR).
* No other life-threatening condition.
* No evidence of sepsis.
* No evidence of superficial skin infection at site of surgery and intervention.
* An established diagnosis of either:

  * cervical myelopathy with modified Japanese Orthopaedic Association score of 8-14, or
  * acute cervical / thoracic SCI with ASIA Impairment Scale grade A-D (as assessed within 72 hours of injury) with neurologic level of injury (NLI) from C2 to T12.
* The ability to undergo, or have had, surgical intervention. -. The ability to undergo transcutaneous intervention including study procedures in the posterior cervical or thoracic midline at or after 14 days from surgery.

Exclusion Criteria:

* Any concomitant impairment of the upper and lower limb at baseline that could potentially confound the neurologic assessments; including but not limited to traumatic or disease conditions like brachial plexus injury, peripheral neuropathy, spinal hematoma, transverse myelitis, non-compressive myelopathy, dementia, and Parkinson's disease.
* mJOA of >= 15 and <= 7, or AIS grade E tSCI at baseline assessment.
* Currently involved in another non-observational ntSCI or tSCI study, or receiving another interventional drug, that could interfere with recordings and confound adverse events.
* Other illness (including mental disorder) that could preclude accurate medical and neurological evaluation, at discretion of the treating surgeon and/or principal investigator.
* Unable to commit to the follow-up schedule.
* Recent history of regular substance abuse (illicit drugs, alcohol), which in the opinion of the investigator would interfere with the subject's participation in the study.
* Any condition likely to result in the patient's death within the next 12 months.
* Prisoner.
* Pregnancy.
* Cardiac pacemaker dependent, unable to undergo electrical stimulation.
* Brain implant, skull prosthesis, plate and screws limiting transcranial stimulation.
* Tattoo at site of skin electrode that causes heat/pain during stimulation.
* Subjects who in the opinion of the investigator are not suitable for inclusion in the study, with reason documented.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) | Twelve Months
  An empirically validated and open worksheet for evaluation of sensation from C2 to S4-5, and motor strength of all major limb myotomes from C5-T1 and L2-S1. This determines the neurologic level of injury (NLI) and severity of motor and sensory completeness, with sensorimotor complete, sensory incomplete, motor incomplete without anti-gravity strength, motor incomplete with anti-gravity strength, and no significant deficit.
ASIA Impairment Scale (ASIA / AIS) | Twelve Months
  The product of the ISNCSCI examination includes a standard motor score (0-5) in five muscle groups in upper and lower extremity bilaterally with total extremity motor score of 100 (5 x [5 upper + 5 lower] x 2).
Modified Japanese Orthopaedic Association (mJOA) | Perioperative
  Validated in cervical myelopathy, the mJOA scale is a patient reported functional scale with 18 points assessing four domains, including: upper extremity (0 - 7), lower extremity (0-7), sensory (0-3), and micturition (0-3). This scale is further divided into severe (</=11), moderate (12-14), and mild (>/=15), with scores <8 reflecting inability to perform clinical assessments (and are excluded).
Blood Pressure | Perioperative
  Systolic and diastolic. Measured in mmHg
Orthostatic Blood Pressure | Perioperative
  As defined by a sustained reduction in systolic blood pressure of at least 20 mmHg or diastolic blood pressure of 10 mmHg within three minutes of standing after being supine for five minutes.
Post-Void Residual | Perioperative
  Defined as the amount of urine remaining in the bladder following urination. Measured in milliliters.
Upper Extremity: Grip Strength | Twelve Months
  Dynamometry measuring grip strength of both hands with participant directed to squeeze a force gauge between their thumb base and fingers at the distal interphalangeal joint. Average of three attempts, measured in kg of force.
GRASSP | Twelve Months
  Gross and fine motor function of the hand is tested with subcomponents while manipulating common, but standardized, objects including jar and water bottle opening, grasping of key, coin, nut and bolt, and nine-peg test. Measured in time (seconds) to completion and/or percentage of completion in a given time period.
Lower Extremity: 10 Meter Walk Test | Twelve Months
  The participant is instructed to walk as fast and accurately as possible across a 10- meter length of hallway, without adaptive devices. This can be consistently recorded whether starting at rest or when already walking 'at speed'. Measured in seconds.
GAITRite Walking Assessment | Twelve Months
  Quantitative analysis of gait using an electronic pressure mat, measured with gait stability ratio (single stance time / double stance time). Measured in time (seconds) and distance (centimeters).
SCIM-vIII (PROM) | Twelve Months
  self-reported questionnaire comprised of 19 questions on daily tasks with a total score between 0 and 100 and subscales for self-care, respiration & sphincter management, and mobility.
WHOQOL-BREF | Twelve Months
  A questionnaire validated in, but not specific to, people with SCI. The WHOQOL-BREF been found to have excellent reliability, adequate-to-excellent validity with complete and incomplete SCI, and acceptable ceiling or floor effects. Measured as a raw score and converted to a percentage with higher values indicating a more positive result.

SECONDARY OUTCOMES:
Adverse Event Rate | Twelve Months
  An adverse event is any undesirable experience associated with the use of a medical product or intervention in a patient. Will be documented as a log and quantified against the number of enrolled participants as a percentage.
Serious Adverse Event Rate | Twelve Months
  A serious adverse event is an adverse event that results in:
  * Death
  * The participant experiencing a substantial risk of dying at the time of the event.
  * Admission to the hospital, or prolongation of hospitalization.
  * Disability, or permanent physical function.
  * Other serious o important medical events as determined by the principal investigator.
  Will be documented as a log and quantified against the number of enrolled participants as a percentage.
Adherence to Protocol | Twelve Months
  Documentation of completion of protocol waypoints (i.e. follow-up visits, intervention steps) expressed as a rate.
Data Collection and Monitoring | Twelve Months
  Documentation of completed data collection waypoints expressed as a rate.

CONTACTS AND LOCATIONS:
Overall Officials: Jared Wilcox, MD, PhD, Principal Investigator — University of Kentucky Neurosurgery
Locations (1):
- University of Kentucky - Chandler Medical Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided